CLINICAL TRIAL: NCT04591808
Title: Efficacy and Safety of Atorvastatin + Perindopril Fixed-Dose Combination S05167 in Adult Patients With Arterial Hypertension and Dyslipidemia, 8 Weeks, Phase 3, Randomized, Double-blind, Active-control, Multinational, Multi-center, Parallel Study
Brief Title: Efficacy and Safety of Atorvastatin + Perindopril Fixed-Dose Combination S05167 in Adult Patients With Arterial Hypertension and Dyslipidemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: for strategic reasons
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL3-05167-005
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Dyslipidemias; Hypertension
Keywords: Dyslipidemia; Hypertension; Cardiovascular; Atorvastatin; Perindopril; HMG-CoA reductase inhibitor; ACE inhibitor; Fixed combination
MeSH Terms: conditions — Dyslipidemias; Hypertension | interventions — Atorvastatin; Perindopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- S05167 (Experimental)
  Interventions: Drug: Atorvastatin/Perindopril
- Lipitor® (Active Comparator)
  Interventions: Drug: Atorvastatin
- Coversyl® (Active Comparator)
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Atorvastatin/Perindopril — 1 over-encapsulated S05167 capsule, fixed dose combination of Atorvastatin/Perindopril Arginine 40/10 mg, will be administered once daily each day before breakfast during 8 weeks.
  Arms: S05167
Drug: Atorvastatin — 1 over-encapsulated atorvastatin 40 mg tablet will be administered once daily each day before breakfast during 8 weeks.
  Arms: Lipitor®
Drug: Perindopril — 1 over-encapsulated perindopril 10 mg tablet will be administered once daily each day before breakfast during 8 weeks.
  Arms: Coversyl®

SUMMARY:
The purpose of this study is to demonstrate the superiority of atorvastatin/perindopril fixed dose combination (FDC) S05167 as compared to atorvastatin reference drug alone or perindopril drug alone on systolic blood pressure decrease and LDL cholesterol decrease respectively in patients presenting with hypertension and dyslipidemia after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women from 18 to 79 years old who can comply with the study requirements and timetable,
2. Patients diagnosed with Essential hypertension (as documented in patient's medical file). The diagnosis of hypertension should be based on at least two BP measurements on at least two visits.

   Uncontrolled hypertensive patients currently under monotherapy treatment within at least 4 weeks (except patients treated by perindopril) for combined systolic and diastolic hypertension (140 mmHg ≤ SBP < 160 mmHg and 90 mmHg ≤ DBP < 100 mmHg).

   or Hypertensive patients naïve of treatment with 150 mmHg ≤ SBP <160 mmHg and 90 mmHg ≤ DBP < 100 mmHg.
3. Dysplipidemic patients: naïve of treatment or uncontrolled with statin at lowest dose within at least 4 weeks with 110 mg/ Decilitre (dL) (or 2.84 millimole [mmol] /L) ≤ LDL-c < 190 mg/dL (or 4.91 mmol/L) according to a previous laboratory result within 12 months.

Exclusion Criteria:

1. Unlikely to cooperate in the study,
2. Pregnant and lactating women,

4. Participation in another study at the same time or having participated in another study within 3 months before selection participation in noninterventional registries or epidemiological studies is allowed,

6.Patients treated with >1 anti-hypertensive drug or >1 Lipid lowering drug,

7.Patients previously treated with atorvastatin and/or perindopril,

8.Known resistance to ACE inhibitors,

9.Patients treated with beta-blockers or alpha-blockers,

10. Patients with liver disease or renal impairment,

11.Certain known cardiovascular diseases or cardiac rhythm disorders,

12.Known or suspected symptomatic orthostatic hypotension,

13.Familial hypercholesterolemia,

14.Secondary hypertension or dyslipidemia,

15.Patients who are hypersensitive to atorvastatin, perindopril or to any of the excipients of study drugs,

16.Hypersensitivity to any other ACE inhibitor,

17.History of angioedema associated with previous ACE inhibitor therapy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | Over 8 weeks
  Mean change from baseline in sitting systolic blood pressure (SBP) in the S05167 group as compared with the Lipitor group (in terms of superiority)
Low-Density Lipoprotein Cholesterol (LDLc) | Over 8 weeks
  Percent of change from baseline in Low-Density Lipoprotein Cholesterol (LDLc) in the S05167 group as compared with the Coversyl group (in terms of superiority)

SECONDARY OUTCOMES:
Systolic blood pressure (SBP) | Over 8 weeks
  Mean change from baseline in sitting systolic blood pressure (SBP) in the S05167 group as compared with Coversyl group
Density Lipoprotein Cholesterol (LDLc) | Over 8 weeks
  Percent of change from baseline in Low-Density Lipoprotein Cholesterol (LDLc) level in the S05167 group as compared with the Lipitor group
Diastolic blood pressure (DBP) | Over 8 weeks
  Mean change from baseline in diastolic blood pressure (DBP) in each group
Pulse Pressure | Over 8 weeks
  Mean change from baseline Pulse Pressure in each group
Lipid parameters | Over 8 weeks
  Percent of Change from baseline
Blood pressure response | Over 8 weeks
  Percent of responders (in terms of blood pressure response defined by patients with BP< 140/90 mm Hg or SBP decrease > = 20 mm Hg or DBP decrease > =10 mm Hg)
Blood pressure control | Over 8 weeks
  Percent of blood pressure control: BP< 140/80 mm Hg AND % of blood pressure control: BP < 130/80 mm Hg
Lipids control | Over 8 weeks
  Percent of responders (in terms of lipids control: an absolute reduction to an LDLc level< 2.6 mmol/L [100 mg/dL] or a reduction at least 50%
Adverse events and Serious adverse events (SAE) | Over 8 weeks
  Emergent Adverse events and Serious adverse events (SAE)
Vital signs | Over 8 weeks
  Blood pressure (BP)
Vital signs | Over 8 weeks
  Pulse rate (PR)
Vital signs | Over 8 weeks
  Respiratory rate (RR)
Electrocardiogram | Over 8 weeks
  Significant abnormalities observed from ECG
Clinical lab tests | Over 8 weeks
  Relevant deviations of laboratory test results

CONTACTS AND LOCATIONS:
Locations (43):
- Georgia (8):
  - LTD "Clinic-LJ", Kutaisi
  - LTD "Marnecore", Marneuli
  - "Aleksandre Aladashvili Clinic" LLC, Tbilisi
  - Israel-Georgian Medical Research Clinic "Helsicore", Tbilisi
  - Bokhua Memorial Cardiovascular Center, Tbilisi
  - Ltd "Digomi Medical Center", Tbilisi
  - LTD "MediClubGeorgia", Tbilisi
  - Emergency Cardiology Center n.a. Acad G Chapidze, Tbilisi
- Russia (22):
  - FSI "Northern Medical Clinical Centre n.a. N.A. Semashko FMBA of Russia", Arkhangelsk
  - Сity clinical hospital #1 named after E.E.Volosevich, Arkhangelsk
  - Non-State Institution of Healthcare "Railway Clinical Hospital at station Chelyabinsk of open joint-stock company "Russian Railways", Chelyabinsk
  - Federal State Institution "National Medical Research Center for Preventive Medicine" of the Ministry of Healthcare of the Russian Federation, Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "City Clinical Hospital No. 17 of the Department of Healthcare of the City of Moscow", Moscow
  - State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital #51" of Department of Healthcare of Moscow, Moscow
  - "Orenburg State Medical University" based on Municipal State healthcare Institution "City Hospital emergency # 1" of the city of Orenburg, Orenburg
  - SBHI "Penza Regional Clinical Hospital n.a. N.N. Burdenko", Penza
  - State budgetary institution "Ryazan' regional clinical hospital", Ryazan
  - Saint Petersburg state budgetary institution of healthcare "City policlinic #109", Saint Petersburg
  - GBOU VPO "North-Western State Medical University named after I.I. Mechnikov" , the department faculty and hospital care, court number 5, Saint Petersburg
  - Medical Research Institute, LLC, Saint Petersburg
  - SPB SBHI "City Hospital # 38 n.a. N.A. Semashko", Saint Petersburg
  - Saint-Petersburg GUZ "City Hospital #40 of the Resort District", Saint Petersburg
  - St. Petersburg State Institution of Health "City Hospital № 15" Cardiology Care Unit, Saint Petersburg
  - St. Petersburg State Budgetary Institution of Healthcare "Diagnostic center #85", Saint Petersburg
  - SPB SBHI "Pokrovskaya City Hospital", Saint Petersburg
  - LLC "MART" Sankt Petersburg, Saint Petersburg
  - Saratov Research Cardiology Institute of Roszdrav, Saratov
  - State Budgetary institutionof heath of Tver region "Region clinical hospital", Tver'
  - State Institution of Healthcare Vladimir region ''City Hospital № 4 of Vladimir ", Vladimir
  - State Budgetary institution of heath of Yaroslavl region "Regional clinical hospital", Yaroslavl
- Ukraine (13):
  - State Higher Educational Institution "Ivano-Frankivsk National Medical University", Chair of Internal Medicine #2 and Nursing based on Communal Institution Ivano-Frankivsk Regional Clinical Cardiological Center, Chronic Ischaemic Heart Disease Department, Ivano-Frankivsk
  - Ivano-Frankivsk central city clinical hospital, Cardiology department, Ivano-Frankivsk
  - "L.T. Malaya Therapy National Institute of the National Institute of Medical Science of Ukraine" Department of aging and prevention of metabolic-associated diseases, Kharkiv
  - The Training and Research Medical Complex "The University Clinic" of the Kharkiv National Medical University, Department of Therapy, National Pharmaceutical University, Chair of Pharmacotherapy, Kharkiv
  - State Institution "Institute of gerontology named after D.F. Chebotaryov НAMS of Ukraine, Department of Clinical and Epidemiological Cardiology, Kiev
  - Medical center ''CONSILIUM MEDICAL'', Kyiv
  - Danylo Halytskyi Lviv National Medical University Department of Therapy No. 1 and Medical Diagnostics of the Faculty of Postgraduate Education, Lviv
  - Chair of Propedeutic of Internal Medicine #1 of Danylo Halytsky Lviv National Medical University based Municipal Non-profit Enterprise "Lviv City Clinical Hospital #5" Out-patient department., Lviv
  - The Medical and Diagnostic Center of LLC "House of Medicine", Odesa
  - Chair of Internal Medicine #3 of Ternopil National Medical University named after I. Gorbachevsky of MOH of Ukraine based on Outpatient Department of Municipal Institution of Ternopil Regional Council "Ternopil University Hospital",, Ternopil
  - Communal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Department of Rheumatology, I. Horbachevsky Ternopil National Medical University of MOH of Ukraine, Chair of Internal Medicine #2, Ternopil
  - Municipal Non-profit Institution "Vinnytsya City Clinical Hospital #1", Therapeutical department; National Pirogov Memorial University, Vinnytsya, Chair of Propedeutics of Internal Medicine;, Vinnytsia
  - Private Small-Scale Enterprise Medical Center "Pulse", Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: [study-level clinical trial data] — https://clinicaltrials.servier.com/